CLINICAL TRIAL: NCT06075810
Title: A Phase 1 Open-Label, First-in-Human Trial of Oral MBQ-167 as Single Agent in Participants With Advanced Breast Cancer
Brief Title: A Study of Oral MBQ-167 in Participants With Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MBQ Pharma (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBQ-ABC001; CDMRP-BC220292 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Breast Neoplasm; Breast Cancer Stage IV
Keywords: Advanced Breast Cancer; Metastatic Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Proto-Oncogene Proteins c-raf; PAK inhibitor MRIA9

STUDY DESIGN:
Intervention Model Description: Open-label dose escalation following a standard 3+3 cohort design with a 21 day Dose Limiting Toxicity (DLT) evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MBQ-167 oral capsule (Experimental): A dose ranging from 10mg to 400mg BID following a standard 3+3 cohort design
  Interventions: Drug: MBQ-167

INTERVENTIONS:
Drug: MBQ-167 — MBQ-167, an inhibitor of Rho GTPases Rac and Cdc42
  Other Names: Rac and Cdc42 inhibitor; Rac inhibitor; Cdc42 inhibitor; PAK inhibitor; Rac/Cdc42 inhibitor

SUMMARY:
A Phase 1, open-label, dose-escalation clinical trial of MBQ-167 in participants with advanced Breast Cancer for whom Standard of Care (SOC) has failed or has proven intolerable.

DETAILED DESCRIPTION:
The main questions this clinical trial aims to answer are:

* What, if any, are the side effects of different dose levels in humans?
* What is the maximum tolerated dose?
* How does the human body process the drug?
* Does the drug slow, stop or eliminate cancer in human participants?

Participants will be asked to:

* provide informed consent
* be evaluated by physicians and provide laboratory specimens to determine if eligible
* take MBQ-167 orally twice a day for at least 21 days
* may continue dosing, if safe to do so, until not effective or other decision to stop is made
* participate in multiple visits that include additional evaluations, laboratory tests and diary review until after stopping the investigational drug

ELIGIBILITY:
Key Inclusion Criteria:

* The investigator will evaluate these and other criteria to determine whether a participant can be included in this study.
* Histologically and/or cytologically confirmed advanced breast cancer which has progressed after treatment with approved therapies or for which there are no standard therapies available.
* Participants with known brain metastases may be eligible if specific conditions are met.
* Life expectancy ≥6 months, in the opinion of the investigator, after starting MBQ-167.
* Are able to swallow capsules twice daily with a meal.

Key Exclusion Criteria:

* The investigator will evaluate these and other criteria to determine whether a participant should be excluded from this study.
* Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the bioavailability of MBQ-167.
* Females who are pregnant or breastfeeding.
* Participants who have received any anticancer treatment within 4 weeks or any investigational agent within 28 days prior to the first dose of trial drug or who have not recovered from any acute toxicity greater than Grade 0 or 1 related to previous anticancer treatment.
* Participants who have received any anticancer treatment within 4 weeks or any investigational agent within 28 days prior to the first dose of trial drug or who have not recovered from any acute toxicity greater than Grade 0 or 1 related to previous anticancer treatment.
* Active malignancies other than advanced breast cancer will be excluded from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 days
  To find the maximum tolerated dose (MTD) of MBQ-167 as a single agent administered orally, BID continuously for 21 days in participants with Advanced Breast Cancer (ABC) by evaluating for the presence or absence of dose-limiting toxicity (DLT) related to MBQ-167 administered in cohorts of participants at escalating sequential cohort dose levels.

SECONDARY OUTCOMES:
MBQ-167 PK parameter (Cmax/min) | 56 days
  Maximum and minimum observed plasma concentration at steady state
MBQ-167 PK parameter (tmax) | 56 days
  Time to maximum plasma concentration
MBQ-167 PK parameter (t1/2) | 56 days
  Terminal elimination half-life
MBQ-167 PK parameter (AUC (0-t,0-24,∞)) | 56 days
  Area under the concentration-time curve over the dosing interval time from time 0
MBQ-167 PD parameter (differential gene expression) | 16 days
  Observed quantitative measurement of gene expression change from baseline
MBQ-167 PK/PD parameter (minimum dose for therapeutic response) | 56 days
  Correlate differential gene expression change, objective response and PK parameter Cmax/min to identify a minimum dose for therapeutic response

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sankar, MD, Study Director — CMO, MBQ Pharma
Locations (4):
- United States (3):
  - Precision Next Gen Oncology & Research Center, Beverly Hills, California
  - Florida Cancer Specialists / Sarah Cannon Research Institute / SCRI, Sarasota, Florida
  - Sarah Cannon Research Institute/SCRI, Nashville, Tennessee
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Collazo A, Ruiz-Calderon JF, Picon H, Borrero-Garcia LD, Lopez I, Castillo-Pichardo L, Del Mar Maldonado M, Duconge J, Medina JI, Bayro MJ, Hernandez-O'Farrill E, Vlaar CP, Dharmawardhane S. Efficacy of Rac and Cdc42 Inhibitor MBQ-167 in Triple-negative Breast Cancer. Mol Cancer Ther. 2021 Dec;20(12):2420-2432. doi: 10.1158/1535-7163.MCT-21-0348. Epub 2021 Oct 4. PMID 34607932
- [Background] Medina JI, Cruz-Collazo A, Del Mar Maldonado M, Gascot TM, Borrero-Garcia LD, Cooke M, Kazanietz MG, O'Farril EH, Vlaar CP, Dharmawardhane S. Characterization of Novel Derivatives of MBQ-167, an inhibitor of the GTP-binding proteins Rac/Cdc42. Cancer Res Commun. 2022 Dec;2(12):1711-1726. doi: 10.1158/2767-9764.crc-22-0303. Epub 2022 Dec 29. PMID 36861094
- [Background] Humphries-Bickley T, Castillo-Pichardo L, Hernandez-O'Farrill E, Borrero-Garcia LD, Forestier-Roman I, Gerena Y, Blanco M, Rivera-Robles MJ, Rodriguez-Medina JR, Cubano LA, Vlaar CP, Dharmawardhane S. Characterization of a Dual Rac/Cdc42 Inhibitor MBQ-167 in Metastatic Cancer. Mol Cancer Ther. 2017 May;16(5):805-818. doi: 10.1158/1535-7163.MCT-16-0442. PMID 28450422
- [Background] Torres-Sanchez A, Rivera-Robles M, Castillo-Pichardo L, Martinez-Ferrer M, Dorta-Estremera SM, Dharmawardhane S. Rac and Cdc42 inhibitors reduce macrophage function in breast cancer preclinical models. Front Oncol. 2023 Jun 16;13:1152458. doi: 10.3389/fonc.2023.1152458. eCollection 2023. PMID 37397366
- [Background] Maldonado MDM, Dharmawardhane S. Targeting Rac and Cdc42 GTPases in Cancer. Cancer Res. 2018 Jun 15;78(12):3101-3111. doi: 10.1158/0008-5472.CAN-18-0619. Epub 2018 Jun 1. PMID 29858187
- [Background] Borrero-Garcia LD, Del Mar Maldonado M, Medina-Velazquez J, Troche-Torres AL, Velazquez L, Grafals-Ruiz N, Dharmawardhane S. Rac inhibition as a novel therapeutic strategy for EGFR/HER2 targeted therapy resistant breast cancer. BMC Cancer. 2021 Jun 1;21(1):652. doi: 10.1186/s12885-021-08366-7. PMID 34074257